CLINICAL TRIAL: NCT07265089
Title: Clinical and Radiographic Evaluation of Success Rate of Zinc Oxide-Ozonated Olive Oil Versus Metapex as Root Canal Filling Materials in Primary Anterior Teeth: Randomized Clinical Trial
Brief Title: Zinc Oxide-Ozonated Olive Oil vs Metapex in Primary Anterior Teeth
Acronym: ZO-OOO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raheeq Babiker Ibrahim Babiker, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-PEDO-ZOO vs MTX
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Carious Anterior Teeth
Keywords: "Zinc Oxide", "Ozonated Olive Oil", "Metapex", "Primary Teeth", "Pulpectomy", "Randomized Clinical Trial".
MeSH Terms: interventions — Metapex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Zinc Oxide-Ozonated Olive Oil (Experimental): Zinc oxide powder will be mixed with ozonated olive oil until a creamy, workable consistency is achieved.
  Interventions: Other: Zinc Oxide-Ozonated Olive Oil
- Group B Metapex (Experimental): Premixed calcium hydroxide with iodoform paste
  Interventions: Other: Metapex

INTERVENTIONS:
Other: Zinc Oxide-Ozonated Olive Oil — Children aged 3-5 years with primary anterior teeth requiring pulpectomy will receive treatment under rubber dam isolation. After achieving local anesthesia, an access cavity will be prepared using sterile round burs with water coolant. Working length will be determined using an apex locator, and biomechanical preparation will be performed with K-files.Irrigation will be done with normal saline and 1% sodium hypochlorite, followed by drying with paper points.
  The canal will then be obturated with a freshly prepared mixture of zinc oxide powder and ozonated olive oil placed using a lentulo spiral, avoiding overfilling. The access cavity will be sealed with glass ionomer and restored with light-cured composite. Follow-up will occur at 3, 6, 9, and 12 months.
  Arms: Group A Zinc Oxide-Ozonated Olive Oil
Other: Metapex — Children aged 3-5 years with primary anterior teeth requiring pulpectomy will receive treatment under rubber dam isolation. After achieving local anesthesia, an access cavity will be prepared using sterile round burs with water coolant. Working length will be determined using an apex locator, and biomechanical preparation will be performed with K-files.and irrigation with normal saline and 1% sodium hypochlorite. After drying, the root canal will be filled with Metapex (premixed calcium hydroxide and iodoform paste) delivered via syringe with a fine tip until proper fill is confirmed radiographically. The canal will then be sealed with glass ionomer and restored with light-cured composite. Follow-up will be performed at 3, 6, 9, and 12 months.
  Arms: Group B Metapex

SUMMARY:
This randomized clinical trial compares zinc oxide-ozonated olive oil and Metapex as root canal filling materials in primary anterior teeth of children aged 3-5 years.

The study aims to evaluate their clinical and radiographic success over 12 months.Clinical evaluation includes pain, swelling, and mobility; radiographic evaluation includes periapical healing and resorption.

DETAILED DESCRIPTION:
Dental caries in primary anterior teeth significantly compromises aesthetics and function, particularly affecting children's psychosocial well-being and oral development. Esthetically, carious lesions in these visible teeth can lead to social avoidance, reduced self-esteem, and bullying risks, as children may avoid smiling or participating in activities. Pulpectomy of primary teeth is a critical to maintain arch integrity, function, and aesthetics in the pediatric population. Zinc oxide eugenol (ZOE) has been the most commonly used filling material in pulptherapy of primary teeth, achieving moderate to high success rates exceeding 90%. However, the slow resorption rate, which may not match the physiological root resorption of primary teeth, potentially leading to delayed natural exfoliation and complications with the eruption of permanent successors. it can also induce necrosis and delayed healing.

(ZOE) can cause irritation and sensitivity when in contact with oral tissues, primarily due to the eugenol component. Eugenol is recognized as a sensitizer and can induce both localized irritation and hypersensitivity reactions, including contact dermatitis, contact stomatitis, and, in rare cases, immediate allergic responses such as urticaria and generalized itching shortly after application.

Olive oil is a vegetal oil it contains antioxidants that enhance properties which can potentially overcome the limited antimicrobial activity of traditional ZOE. Ozonated olive oil has demonstrated excellent biocompatibility with surrounding tissues. This reduces the adverse reactions or irritation, making it a safer alternative for pediatric patients. Zinc oxide-ozonated olive oil may reduce the chances of overfilling and subsequent eruption complications. Promotes tissue repair and healing due to its anti-inflammatory and regenerative properties. This can contribute to quicker recovery and better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3-5 years.
2. Primary anterior teeth requiring root canal treatment due to irreversible pulpitis.
3. Cooperative behavior child.
4. Parents provided written informed consent. -

Exclusion Criteria:

1. Medically compromised children.
2. Tooth with advanced root resorption.
3. Non-restorable crown structures.
4. Tooth with abscess or fistula.
5. Allergies or hypersensitivity to any of the materials used e.g., zinc oxide, olive oil, or calcium hydroxide and Idoform (components of Metapex).
6. Unable to attend follow-up visits.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success: absence of pain, swelling, tenderness, or mobility | 12 month intervals T0: 0 T1: 3month T2: 6month T3: 9month T4: 12month

SECONDARY OUTCOMES:
Radiographic success: absence of periapical radiolucency or root resorption | 12 month intervals T0:0 T2: 6 month T4: 12month

CONTACTS AND LOCATIONS:
Overall Officials: Adel Elbardissy Professor of Pediatric Dentistry and Dental Public Health, Prof. Doctor, Study Director — Faculty of Dentistry, Cairo University, Egypt
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No